CLINICAL TRIAL: NCT00443690
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Effects of KW-3902 Injectable Emulsion on Heart Failure Signs and Symptoms, Diuresis, Renal Function, and Clinical Outcomes in Subjects Hospitalized With Worsening Renal Function and Heart Failure Requiring Intravenous Therapy
Brief Title: Placebo-Controlled Randomized Study of KW-3902 for Subjects Hospitalized With Worsening Renal Function and Heart Failure Requiring IV Therapy
Acronym: REACH UP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovaCardia, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKI-303; 2007_805; MK7418-303
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure; diuretic; renal impairment; renal function
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — rolofylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): placebo control
  Interventions: Drug: Comparator: Placebo (unspecified)
- 1 (Experimental): KW-3902IV
  Interventions: Drug: rolofylline

INTERVENTIONS:
Drug: rolofylline — rolofylline 30 mg IV QD; 3 days
  Other Names: KW-3902IV; MK7418
  Arms: 1
Drug: Comparator: Placebo (unspecified) — rolofylline Pbo 30 mg IV QD; 3 days
  Arms: 2

SUMMARY:
To evaluate the effect of KW-3902IV, in addition to standard therapy, on the proportion of worsening heart failure and worsening renal function, and on the proportion of deaths or rehospitalizations for heart failure or worsening renal function, and to estimate and compare within-trial medical resource utilization and direct medical costs between subjects treated with KW 3902IV versus placebo.

DETAILED DESCRIPTION:
Loop diuretics are generally first line therapy in patients hospitalized with acute heart failure syndrome (AHFS). Their use far exceeds that of vasoactive agents. Tubuloglomerular feedback (TGF) is the body's compensatory response to avoid excess fluid loss, and it is activated when elevated sodium concentrations in the distal tubule are detected. TGF is proposed as a contributing factor for the observed diuretic resistance that occurs in patients with heart failure. Higher doses of diuretics are required to overcome the decreased natriuresis and reduced RBF induced by TGF. Ultimately, this action creates a vicious cycle of worsening renal function and diminished diuretic effectiveness.

The primary pharmacologic rationale for the use of KW-3902 in subjects with AHFS is its mechanism of action as an adenosine A1 receptor antagonist. TGF promotes release of adenosine, and adenosine binding to A1 receptors causes vasoconstriction of the afferent arteriole, decreased RBF, and enhanced sodium reabsorption by the proximal tubule. This action results in a decrease in GFR, diminished renal function, and sodium and water retention. Blocking adenosine A1 receptors via a selective adenosine receptor antagonist may limit sodium reabsorption by the proximal tubules without triggering TGF. It promotes vasodilation of the afferent arteriole of the glomerulus, and thus, this strategy offers the potential to overcome diuretic resistance or enhance diuretic responsiveness. It may also reduce the need for increasing diuretic doses that have been associated with worse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea at rest or with minimal exertion at randomization
* Fluid overload
* Estimated creatinine clearance (CrCl) between 20-60 mL/min
* Worsening renal function
* Anticipated need for IV diuretic treatment for at least 48 hours after the start of study drug
* BNP >500 pg/mL or NT-pro-BNP >2000 pg/mL
* Systolic blood pressure ≥90 mmHg at randomization

Exclusion Criteria:

* IV radiographic contrast within 14 days
* IV vasodilators within 6 hours
* Serum potassium <3.5 meq/L
* Ongoing or planned therapy for heart failure with mechanical circulatory or ventilatory support
* Ongoing or planned treatment with ultrafiltration, hemofiltration, or dialysis
* Rapidly progressive acute renal failure
* Evidence of acute tubular necrosis or post-obstructive nephropathy or other exogenous causes of acute kidney injury, unrelated to heart failure
* Severe pulmonary disease
* Significant stenotic mitral or aortic valvular disease
* Heart transplant recipient or admitted for cardiac transplantation or LVAD surgery
* Any major surgery within 2 weeks prior
* evidence of acute coronary syndrome in the 2 weeks prior
* Hgb <8 g/dL, Hct <25%, or active bleeding requiring transfusion
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy.
* Known hepatic impairment
* Non-cardiac pulmonary edema
* Temperature >38°C
* Sepsis or active infection requiring IV anti-microbial treatment
* Administration of an investigational drug or device within 30 days
* Current or anticipated therapy with atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, or voriconazole
* Administration of any vasopressor or inotropic drug within 72 hours
* History of seizure (except febrile seizure)
* Stroke within 2 years
* History of brain tumor of any etiology
* Brain surgery within 2 years
* Encephalitis/meningitis within 2 years
* History of penetrating head trauma
* Closed head injury with loss of consciousness (LOC) over 30 minutes within 2 years
* History of or at risk for alcohol withdrawal seizures
* Advanced Alzheimer's disease
* Advanced multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Effect on heart failure signs and symptoms | through day 7
Effect on renal function | through Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Barry Massie, MD, Study Chair — University of California San Francisco, USA; Christopher O'Connor, MD, Study Chair — Duke University, USA